CLINICAL TRIAL: NCT03604861
Title: Remission From Chronic Opioid Use: Studying Environmental and SocioEconomic Factors on Recovery-The RECOVER Study®
Brief Title: An Observational Study of Environmental and SocioEconomic Factors in Opioid Recovery
Acronym: RECOVER®
Status: Completed | Type: Observational
Sponsor: Indivior Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: INDV-6000-N01
Record Dates: First submitted 2018-07-09; First posted 2018-07-30 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Opioid-use Disorder; Opioid-related Disorders
Keywords: Opioid recovery; Recovery; Opioid-related disorders; Substance-related disorders; Heroin dependence; Opioid dependence; Addiction; Buprenorphine; Opiate substitution treatment; Analgesics; Opioid; Narcotics; Patient outcome assessment; Patient-centered care; Cost of illness; Employment; Health-related quality-of-life; Family relations; Lifestyle; Citizenship
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders; Heroin Dependence; Behavior, Addictive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Not applicable - no defined intervention — Participants who received at least one injection of RBP-6000 or placebo and either withdrew from or completed the Phase III clinical program which included studies NCT02357901 (RB-US-13-0001) and NCT02510014 (RB-US-13-0003) were eligible for the RECOVER Study.

SUMMARY:
The RECOVER Study will examine clinical, environmental and socioeconomic factors in recovery from opioid use disorder (OUD) over a 24-month period following exit from a Phase III clinical program for a buprenorphine extended-release injection (RBP-6000). The study population will consist of participants from studies NCT02357901 (RB-US-13-0001) and NCT02510014 (RB-US-13-0003).

The RECOVER study will characterize OUD subjects' recovery process as they transition from the controlled clinical trial environment to the real world setting.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who received at least one injection in RBP-6000 or placebo in the Phase III clinical program which includes study protocols NCT02357901 (RB-US-13-0001) and NCT02510014 (RB-US-13-0003) and either withdrew from or completed these studies.
* Ability to comply with study protocol requirements for data collection and provide informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are currently diagnosed with moderate or severe OUD according to Diagnostic and Statistical Manual 5 (DSM-5) criteria and for 3 months immediately prior to signing the informed consent form for protocols NCT02357901 (RB-US-13-0001) and/or NCT02510014 (RB-US-13-0003).
Sampling Method: Non-Probability Sample
Enrollment: 534 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Who Reported Abstinent From Opioids For the Previous 7 Days and Previous 28 Days at Month 24 | Month 24
  Based on self-reported abstinence from opioids using the National Survey on Drug Use and Health (NSDUH).
Change from Baseline in Percentage of Participants Who Reported Abstinent From Opioids For the Previous 7 Days At Months 3, 6, 9, 12, 15, 18, 21, 24 | Baseline (Day 1), Months 3, 6, 9, 12, 15, 18, 21, 24
  Based on self-reported abstinence from opioids using the National Survey on Drug Use and Health (NSDUH).
Change from Baseline in Percentage of Participants Who Reported Abstinent From Opioids For the Previous 28 Days At Months 3, 6, 9, 12, 15, 18, 21, 24 | Baseline (Day 1), Months 3, 6, 9, 12, 15, 18, 21, 24
  Based on self-reported abstinence from opioids using the National Survey on Drug Use and Health (NSDUH).
Percentage of Participants Who Reported Abstinent From Opioids For the Previous 7 Days and Confirmed by Urine Drug Screen (UDS) at Month 24 | Month 24
  Based on self-reported abstinence from opioids (using NSDUH), and confirmed by UDS.
Change from Baseline in Percentage of Participants Who Reported Abstinent From Opioids For the Previous 7 Days and Confirmed by UDS At Months 3, 6, 9, 12, 15, 18, 21, 24 | Baseline (Day 1), Months 3, 6, 9, 12, 15, 18, 21, 24
  Based on self-reported abstinence from opioids (using NSDUH), and confirmed by UDS.

OTHER OUTCOMES:
Change from Baseline in 12-Item Short Form Health Survey, Version 2 (SF-12v2) to Months 12 and 24 | Baseline (Day 1), Months 12 and 24
Change from Baseline in the Subjective Opioid Withdrawal Scale (SOWS) to Months 12 and 24 | Baseline (Day 1), Months 12 and 24
Change from Baseline in the Beck Depression Inventory (BDI) to Months 12 and 24 | Baseline (Day 1), Months 12 and 24
Change from Baseline in the Brief Pain Inventory (BPI) to Months 12 and 24 | Baseline (Day 1), Months 12 and 24
Percentage of Participants Currently Employed at Baseline, Month 12 and Month 24 | Baseline (Day 1), Months 12 and 24
Amount of Health Care Resource Utilization (HCRU) at Months 1-12 and Months 13-24 | Months 1-12 and Months 13-24
  HCRU information includes hospitalizations, residential substance abuse treatment, general practitioner/specialist/and counseling visits, and emergency department (ED) visits.
Number of Crimes Committed at Baseline, Months 1-12 and Months 13-24 | Baseline (Months -6 to Day 1), Months 1-12 and Months 13-24
  Participants complete surveys to identify the number and type of criminal incidents in a given time frame. These questions include information on arrests, violence, unlawful behaviors, and driver's license status.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Global Medicines Development, Study Chair — Indivior Inc.
Locations (35):
- United States (35):
  - Winston Technology Research LLC, Haleyville, Alabama
  - Boyett Health Services, Hamilton, Alabama
  - Woodland International Research Group, Little Rock, Arkansas
  - Behavioral Research Specialists, Glendale, California
  - Collaborative Neuroscience Networks, Inc., Long Beach, California
  - Synergy Research Center, National City, California
  - North County Clinical Research, Oceanside, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Amit Vijapura, Jacksonville, Florida
  - Meridien Research, Lakeland, Florida
  - Try Research, Maitland, Florida
  - Innovative Clinical Research, Miami, Florida
  - Scientific Clinical Research, Miami, Florida
  - Research Centers of America, Oakland Park, Florida
  - Louisiana Research Associates, New Orleans, Louisiana
  - Louisiana Clinical Research, Shreveport, Louisiana
  - Stanley Street Treatment and Resources, Fall River, Massachusetts
  - Adams Clinical Trials, Watertown, Massachusetts
  - Precise Research Centers, Inc., Flowood, Mississippi
  - St. Louis Clinical Trials, St Louis, Missouri
  - Altea Research Institute, Las Vegas, Nevada
  - Hassman Research Institute, Berlin, New Jersey
  - Center for Emotional Fitness, Cherry Hill, New Jersey
  - The Medical Research Network, LLC, New York, New York
  - Neuro-behavioral Clinical Research, Canton, Ohio
  - Midwest Clinical Research Center, Dayton, Ohio
  - Charak Clinical Research Center, Garfield Heights, Ohio
  - Oklahoma Clinical Research Center, Oklahoma City, Oklahoma
  - Pahl Pharmaceutical Professionals, Oklahoma City, Oklahoma
  - CODA, Portland, Oregon
  - Tipton Medical and Diagnostic Center aka Clinical Research Associates of Central PA, Altoona, Pennsylvania
  - UPenn Treatment Research Center, Philadelphia, Pennsylvania
  - Carolina Clinical Trials, Charleston, South Carolina
  - Pillar Clinic Research, LLC, Dallas, Texas
  - InSite Clinical Research, DeSoto, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Craft WH, Tegge AN, Keith DR, Shin H, Williams J, Athamneh LN, Stein JS, Chilcoat HD, Le Moigne A, DeVeaugh-Geiss A, Bickel WK. Recovery from opioid use disorder: A 4-year post-clinical trial outcomes study. Drug Alcohol Depend. 2022 May 1;234:109389. doi: 10.1016/j.drugalcdep.2022.109389. Epub 2022 Mar 9. PMID 35287034
- [Derived] Ling W, Nadipelli VR, Aldridge AP, Ronquest NA, Solem CT, Chilcoat H, Albright V, Johnson C, Learned SM, Mehra V, Heidbreder C. Recovery From Opioid Use Disorder (OUD) After Monthly Long-acting Buprenorphine Treatment: 12-Month Longitudinal Outcomes From RECOVER, an Observational Study. J Addict Med. 2020 Sep/Oct;14(5):e233-e240. doi: 10.1097/ADM.0000000000000647. PMID 32187112